CLINICAL TRIAL: NCT02336568
Title: The Effect of 21-Days Intranasal Oxytocin on Clinical Symptoms and Social Function in Patients With Post Traumatic Stress Disorder (PTSD), a Randomized Controled Trail
Brief Title: The Effect of 21-Days Intranasal Oxytocin on Patients With Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 370-14CTIL
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: PTSD
Keywords: PTSD, Oxytocin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): intervention: Oxytoine treatments - 20 PTSD patients
  Interventions: Drug: Oxytoine
- Placebo treatments (Placebo Comparator): Other: Placebo treatments- 20 PTSD patients
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Oxytoine — In the first week 24 IU * 2/day. in the 2nd & 3rd 40 IU * 2/day
  Other Names: syntocinon nasal spray nasal
  Arms: intervention
Drug: PLACEBO — In the first week 24 IU * 2/day. in the 2nd & 3rd 40 IU * 2/day
  Arms: Placebo treatments

SUMMARY:
Oxytocin (OT) - a neurohormone and neuromodulator which is mainly synthesized in the hypothalamus - is a mediator stress regulation and improves social bonding. Recently, several theoretical studies suggested that PTSD patients have abnormal functioning of the OT system. According to these theories, dysfunction in the oxytocin system may modulate the interpersonal impairment that characterizes PTSD, and therefore intranasal OT may potentially relieve these symptoms. In two current studies that were conducted in Rambam health care we found that a single dose of intranasal OT reduces anxiety and irritability symptoms, and enhances emotional empathy and compassion, in patients with PTSD. The main goal of this study is to examine the effects of 21-days intranasal Oxytocin on clinical symptoms and social function in these patients.

DETAILED DESCRIPTION:
This study will examine the effect is of 21-days intranasal Oxytocin on clinical symptoms and social function in these patients, in a double blind (treatment/placebo) study design.

ELIGIBILITY:
Inclusion Criteria:

* PTSD patients (DSM-IV criteria)
* Ability to provide written informed consent

Exclusion Criteria:

* Suicidality
* Psychosis
* Borderline Personality
* Arrhythmia
* Cardiac disease (arrythmia, heart failure)
* Hyponatremia
* Hypertension
* Severe renal insufficiency
* Liver cirrhosis
* Lactating or pregnant women, or undergoing fertility treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interviews (CAPS)and self-report questionnaires that examine the symptoms of the disorder and related symptoms (social function and aggressive behavior) | 3 weeks